CLINICAL TRIAL: NCT01540838
Title: Slow Initial β-lactam Infusion With High-dose Paracetamol to Improve the Outcomes of Childhood Bacterial Meningitis, Especially of Pneumococcal Meningitis, in Angola.
Brief Title: Slow Initial β-lactam Infusion With High-dose Paracetamol to Improve the Outcomes of Childhood Bacterial Meningitis
Acronym: INFU/PARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Foundation for Paediatric Research, Finland (Other)
Responsible Party: Principal Investigator, Heikki Peltola, MD, PhD, Profesor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INFU/PARA-BOLU/PLACE
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Meningitis
Keywords: Bacterial meningitis; infusion; bolus; paracetamol
MeSH Terms: conditions — Meningitis, Bacterial | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion with paracetamol (Experimental): Cefotaxime is administered as 12 hourly infusions, together with high dose paracetamol (acetaminophen)
  Interventions: Drug: Infusion with paracetamol
- Bolus with placebo (Active Comparator): Cefotaxime is administered as bolus q.i.d. with a placebo of paracetamol
  Interventions: Drug: Bolus without paracetamol

INTERVENTIONS:
Drug: Infusion with paracetamol — The administration of 250 mg/kg/24 hours cefotaxime during the first 4 days as continuous intravenous infusion, each single infusion lasting for 12 hours (to prevent degradation of the agent), combined with high-dose paracetamol orally; the first dose is 30 mg/kg, then 20 mg/kg every 6 hours for 4 full days.
  Other Names: paracetamol=acetaminophen
  Arms: Infusion with paracetamol
Drug: Bolus without paracetamol — The control intervention consists of 250 mg/kg/24 hours cefotaxime administered traditionally with intermittent i.v. boluses and the place bo of paracetamol orally, both repeated every 6 hours (qid) for 4 days.
  Other Names: Paracetamol=acetaminophen
  Arms: Bolus with placebo

SUMMARY:
The main purpose of this trial is to test if mortality of childhood bacterial meningitis can be reduced by slow, continuous infusion of cefotaxime initially, instead of the traditional bolus administration four times daily (qid), combined with high-dose paracetamol orally, when both treatments are executed for the first 4 days. The series will be collected at Hospital Pediátrico David Bernardino, Luanda, Angola.

The recruitment of patients begins, the conditions permitting, in early 2012. The criteria for patient participation is a child at the age of 2 months to 15 years who presents with the symptoms and signs suggestive of bacterial meningitis, for whom a lumbar puncture is performed, and the cerebrospinal fluid analysis suggests bacterial meningitis.

DETAILED DESCRIPTION:
The principal objective of the study is to examine if mortality of childhood bacterial meningitis can be reduced by slow continuous infusion of cefotaxime combined with high-dose paracetamol orally for the first 4 days (instead of the traditional qid administration of cefotaxime without concomitant paracetamol). Children qualifying for entry (see criteria below), whose guardian has given informed consent,will be randomized into 2 treatment arms (see details below)and receive the treatments in a double blind fashion (see details below). Primary and secondary outcomes (detailed below) will be evaluated according to predefined criteria and time points (see below).

Results will be analyzed for all patients in ITT datasets and in prespecified subgroups (etiology, nutritional status, etc.) in both crude and adjusted analysis. The efficacy results will be expressed as OR with 95% confidence intervals.

ELIGIBILITY:
Eligibility criteria:

The study entry is assessed for all children at age 2 months - 15 years who present at these centers with the symptoms and signs suggestive of bacterial meningitis (BM), and to whom lumbar puncture is performed.

Inclusion criteria:

All patients whose cerebrospinal fluid (CSF) turns out to be cloudy, positive by Gram staining or latex agglutination, or shows at least 50 leukocytes per mm3, will be enrolled in the study.

Participants: Exclusion criteria

Exclusion criteria:

1. Trauma, or relevant underlying illness such as intracranial shunt, previous neurological abnormality (cerebral palsy, Down's syndrome, meningitis)
2. Previous hearing impairment (if known)
3. Immunosuppression, except HIV infection
4. More than one parenteral dose of a pretreatment antimicrobial. Children with oral antimicrobials are included, this information being marked in the FOLLOW-UP sheet.
5. Active tuberculosis (if tuberculotic meningitis is diagnosed during trial, it will be included in intention-to-treat (ITT) analysis)
6. Known hepatic disease.

Ages: 2 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki O Peltola, MD, PhD, Study Director — Childrens Hospital of Helsinki University Central Hospital
Locations (1):
- Hospital Pediatrico David Bernardino, Luanda, Angola

IPD SHARING:
Plan to Share IPD: Undecided
We are working on an agreement to share data with all the participants,

REFERENCES:
- [Background] Pelkonen T, Roine I, Cruzeiro ML, Pitkaranta A, Kataja M, Peltola H. Slow initial beta-lactam infusion and oral paracetamol to treat childhood bacterial meningitis: a randomised, controlled trial. Lancet Infect Dis. 2011 Aug;11(8):613-21. doi: 10.1016/S1473-3099(11)70055-X. Epub 2011 May 5. PMID 21550313
- [Derived] Pelkonen T, Roine I, Kallio M, Jahnukainen K, Peltola H. Prevalence and significance of anaemia in childhood bacterial meningitis: a secondary analysis of prospectively collected data from clinical trials in Finland, Latin America and Angola. BMJ Open. 2022 Mar 14;12(3):e057285. doi: 10.1136/bmjopen-2021-057285. PMID 35288394
- [Derived] Savonius O, Rugemalira E, Roine I, Cruzeiro ML, Peltola H, Pelkonen T. Extended Continuous beta-Lactam Infusion With Oral Acetaminophen in Childhood Bacterial Meningitis: A Randomized, Double-blind Clinical Trial. Clin Infect Dis. 2021 May 18;72(10):1738-1744. doi: 10.1093/cid/ciaa341. PMID 32246138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1128 patients were assessed for eligibility at the Hospital´s Emergency Service from Jan 2012 to Jan 2017.
  753 were excluded and 375 enrolled and randomized.
Period: Overall Study
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Started | 188 | 187
Completed | 166 | 164
Not Completed | 22 | 23
Not completed — Open nasogastric tube | 9 | 7
Not completed — Treatment doses missing | 8 | 12
Not completed — Additional antibiotic treatment | 1 | 2
Not completed — Died before treatment initiation | 1 | 1
Not completed — Not BM. Other treatment | 3 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Infusion With Paracetamol | Bolus With Placebo | Total
Number analyzed (Participants) | 188 | 187 | 375
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: The exact age of one patient was unknown.
  months
    number analyzed (Participants) | 187 | 187 | 374
    (all) | 43.6 (42.0) | 45.7 (43.8) | 44.6 (42.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 71 | 158
  Male | 101 | 116 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 188 | 187 | 375
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 179 | 178 | 357
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Angola | 188 | 187 | 375
Weight-for-age, Z-score [Mean (Standard Deviation); unit: Z-score] — The Weight-for-age Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population. These data were calculated using the World Health Organisation (WHO) reference data. Population: Information on the exact age in months was missing from one patient, and the information on the exact weight was missing from one patient.
  Z-score
    number analyzed (Participants) | 187 | 186 | 373
    (all) | -1.179 (1.376) | -1.239 (1.426) | -1.209 (1.400)

OUTCOME MEASURES:

1. Primary Outcome: Day 7 Mortality
Description: All patients who had received at least one dose of treatment and were dead on day 7 from the institution of treatment on day 1.
Time Frame: On day 7 from the institution of treatment
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 187 | 186
Participants | 61 | 64

2. Secondary Outcome: All Deaths During Hospital Stay
Description: All patients who had received at least one dose of treatment and died during the hospital stay.
Time Frame: The outcome was assessed each day until the patient was discharged from the hospital. The longest hospital stay was 84 days, while the last death occurred 39 days after treatment initiation.
Population: All patients who had received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 187 | 186
Participants | 71 | 75

3. Secondary Outcome: Status on the Modified Glasgow Outcome Scale
Description: Scores on the modified Glasgow Outcome Scale which range from a maximum of 5 (best) to a minimum of 1 (worst) points.
  The Glasgow Outcome Scale categorizes the outcome after brain injury into five categories, based on the level and severeness of disability. As hearing impairment is one of the most common sequelae of bacterial meningitis, an assessment of hearing should be included when estimating the grade of disability.
  Hearing thresholds (in decibel, dB) were determined by brainstem evoked response audiometry (BERA), for each ear separately.
Time Frame: Examined at discharge from hospital, except for hearing evaluations which were performed at earliest seven days since the institution of treatment, during the hospital stay. The longest hospital stay was 84 days.
Population: We were finally able to perform post-treatment audiological examinations in solely 37 participants, of whom one lacked information on the neurological outcome. Thus, the Glasgow Outcome Scale score could be estimated for 36 participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 19 | 17
score on a scale | 5 [3 to 5] | 5 [5 to 5]

4. Secondary Outcome: Death or Any Neurological Sequelae on Day 7
Description: Defined as death or any severe neurological sequelae, or hemi- or monoparesis, or ataxia, or psychomotor retardation of any degree.
Time Frame: Examined on day 7 since institution of treatment.
Population: All patients who had received at least one dose of treatment, and from whom the information on any neurological sequelae was available on day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 166 | 168
Participants | 96 | 86

5. Secondary Outcome: A Change in Hearing Threshold Compared to the First Test Result
Description: Hearing thresholds (in decibel, dB) were determined by brainstem evoked response audiometry (BERA), for each ear separately. The better ear's hearing threshold, obtained on admission or shortly thereafter, was compared with the better ear's hearing threshold obtained at earliest after one week of treatment.
Time Frame: Hearing thresholds obtained during any of the first three days after hospital admission were compared with hearing thresholds obtained on day seven or later, during the hospital stay. The longest hospital stay was 84 days.
Population: We were finally able to perform post-treatment audiological examinations in solely 37 participants, and 10 of these lacked primary audiological examinations. Thus, this outcome is reported for 27 participants.
Measure: Median (Inter-Quartile Range); unit: dB
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 13 | 14
dB | 0 [-20 to 0] | 0 [0 to 0]

6. Secondary Outcome: Death or Severe Neurological Sequelae on Day 7
Description: Death or severe neurological sequelae, defined as blindness, tetraplegia/paresis, hydrocephalus requiring a shunt and severe psychomotor retardation
Time Frame: Examined on day 7 since institution of treatment
Population: All patients who received at least one dose of treatment, and of whom information on severe neurological sequelae was available on day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 172 | 173
Participants | 80 | 75

7. Secondary Outcome: Number of Participants With Deafness
Description: Hearing thresholds (in decibel, dB) were determined by brainstem evoked response audiometry (BERA), for each ear separately. Deafness was defined as a hearing threshold >80 dB in the better ear.
Time Frame: This outcome includes hearing thresholds determined at earliest seven days after the institution of treatment, during the hospital stay. The longest hospital stay was 84 days.
Population: We were finally able to perform post-treatment audiological examinations in solely 37 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 20 | 17
Participants | 3 | 1

8. Secondary Outcome: Death or Any Neurological Sequelae at Discharge From Hospital.
Description: as for outcome 4
Time Frame: Examined at discharge from hospital. The longest hospital stay was 84 days.
Population: All patients who hade received at least one dose of treatment, and of whom information on any neurological sequelae was available at discharge from hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 181 | 179
Participants | 104 | 89

9. Secondary Outcome: Death or Severe Neurological Sequelae at Discharge
Description: as for outcome 6
Time Frame: Examined at discharge from hospital. The longest hospital stay was 84 days.
Population: All patients who received at least one dose of treatment, and of whom information on severe neurological sequelae was available at discharge from hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
Number analyzed (Participants) | 186 | 183
Participants | 90 | 85

ADVERSE EVENTS:
Time Frame: During the patient´s hospital stay of at least 7 days until discharge. The longest hospital stay was 84 days.
Description: No specific events or findings, a part from the follow up-data detailed in the protocol, were considered as potential adverse events to be registered because both death, serious sequelae, and/or prolonged hospital stay, given as examples of severe adverse events, are part of the possible course of childhood bacterial meningitis, as such.
  Deaths and other follow-up data were assessed by attending physician.
Arm/Group | Infusion With Paracetamol | Bolus With Placebo
All-Cause Mortality (participants affected / at risk) | 72/188 | 76/187
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/187
Other Adverse Events (participants affected / at risk) | 0/188 | 0/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion With Paracetamol (N=188) | Bolus With Placebo (N=187)
Any adverse events (Nervous system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT01540838/Prot_SAP_000.pdf